CLINICAL TRIAL: NCT02333682
Title: The Response of Serum 25-hydroxyvitamin D to Different Doses of Calcifediol Hy.D Compared to Vitamin D3 Supplementation: A Randomized, Controlled, Double Blind, Long Term Pharmacokinetic Study
Brief Title: Pharmacokinetics of Calcifediol and Cholecalciferol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Leatherhead Food Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-04-17-HDPK; 127927 (Other: Leatherhead Food Research)
Record Dates: First submitted 2014-10-20; First posted 2015-01-07 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Calcifediol; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 25(OH)D3 (Calcifediol Hy.D) 10 mcg (Experimental): 25(OH)D3 (Calcifediol Hy.D), Dose: 10 mcg, 1 capsule/day before breakfast, Duration: 6 months
  Interventions: Dietary Supplement: 25(OH)D3 (Calcifediol Hy.D) 10 mcg
- 25(OH)D3 (Calcifediol Hy.D) 15 mcg (Experimental): 25(OH)D3 (Calcifediol Hy.D), Dose: 15 mcg, 1 capsule/day before breakfast, Duration: 6 months
  Interventions: Dietary Supplement: 25(OH)D3 (Calcifediol Hy.D) 15 mcg
- 25(OH)D3 (Calcifediol Hy.D) 20 mcg (Experimental): 25(OH)D3 (Calcifediol Hy.D), Dose: 20 mcg, 1 capsule/day before breakfast, Duration: 6 months
  Interventions: Dietary Supplement: 25(OH)D3 (Calcifediol Hy.D) 20 mcg
- Vitamin D3 (Cholecalciferol) 20 mcg (Active Comparator): Vitamin D3 (Cholecalciferol), Dose: 20 mcg, 1 capsule/day before breakfast, Duration: 6 months
  Interventions: Dietary Supplement: Vitamin D3 (Cholecalciferol) 20 mcg

INTERVENTIONS:
Dietary Supplement: 25(OH)D3 (Calcifediol Hy.D) 10 mcg — 25(OH)D3 (Calcifediol Hy.D)
  Arms: 25(OH)D3 (Calcifediol Hy.D) 10 mcg
Dietary Supplement: 25(OH)D3 (Calcifediol Hy.D) 15 mcg — 25(OH)D3 (Calcifediol Hy.D)
  Arms: 25(OH)D3 (Calcifediol Hy.D) 15 mcg
Dietary Supplement: 25(OH)D3 (Calcifediol Hy.D) 20 mcg — 25(OH)D3 (Calcifediol Hy.D)
  Arms: 25(OH)D3 (Calcifediol Hy.D) 20 mcg
Dietary Supplement: Vitamin D3 (Cholecalciferol) 20 mcg — Vitamin D3 (Cholecalciferol)
  Arms: Vitamin D3 (Cholecalciferol) 20 mcg

SUMMARY:
The investigators are intending to perform a clinical study in healthy subjects on the pharmacokinetics of different doses of Hy.D Calcifediol compared to vitamin D3 (cholecalciferol) in order to gain insight into the dose response relationship and to assess kinetic differences including the steady state. The metabolites 1,25(OH)2D, 24,25(OH)2D will be assessed throughout the study to assess the metabolism of vitamin D vs. 25(OH)D. Vitamin D3 will be measured throughout the study to assess compliance with the restriction of exogenous vitamin D supplementation.

DETAILED DESCRIPTION:
Reaching consistent levels of 25(OH)D has been shown to be crucial in decreasing falls, fractures and increasing calcium absorption. One way to circumvent the variability of 25(OH)D response to vitamin D might be to use calcifediol supplementation and bypass the 25-hydroxylase enzyme entirely. This approach also permits the physician to achieve desired serum levels in a matter of just a few days, rather than the several weeks required when using native vitamin D. Compared to native vitamin D, calcifediol is more water soluble, has a shorter half-life and increases 25(OH)D levels more quickly. Calcifediol is also more potent, about 3.5 times more potent in raising 25(OH)D levels than vitamin D. Its water solubility may also confer an advantage in patients who have difficulty absorbing fat soluble vitamins. This form of vitamin D metabolite has been used historically to increase calcium absorption, treat osteomalacia, and increase Bone Mineral Density (BMD). Using calcifediol seems to be a practical solution, but little is known about the dose response variability in humans and how it compares to that of native vitamin D. The investigators are intending to perform a clinical study in healthy subjects on the pharmacokinetics of different doses of Hy.D Calcifediol compared to vitamin D3 (cholecalciferol) in order to gain insight into the dose response relationship and to assess kinetic differences including the steady state. The metabolites 1,25(OH)2D, 24,25(OH)2D will be assessed throughout the study to assess the metabolism of vitamin D vs. 25(OH)D. Vitamin D3 will be measured throughout the study to assess compliance with the restriction of exogenous vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males >50 years in age
* Healthy postmenopausal women >50 years in age, who have not experienced a menstrual bleeding for a minimum of 12 months
* BMI between 20-32 kg/m2
* Subject understands the study procedures and signs the informed consent to participate in the study
* Subject has clear understanding of the English language
* Caucasian ethnicity
* Willingness to avoid direct sun exposure and to restrict travel to sunny climates during the whole study period.

Exclusion Criteria:

* Subject has any health conditions that would prevent him/her from fulfilling the study requirements, put the subject at risk or would confound the interpretation of the study results as judged by the Principal Investigator
* Subjects with a history of hypercalcemia (Serum calcium adjusted for albumin of > 2.6 nmol/l)
* Supplemental calcium intake beyond 500 mg per day during the entire study and follow up
* Any vitamin D supplementation within 2 months before the baseline blood draw and during the entire study and follow up
* Subject has gastrointestinal malabsorption (from coeliac disease, colitis, surgery etc.)
* Subject has kidney disease or liver disease
* Medication: Bisphosphonate or Parathyroid Hormone (PTH) treatment, use of steroids in any form, anticonvulsants, antibiotics, antipsychotics, use of any drug that alters fat absorption, e.g. Xenical (Ali).
* Use of Hormone Replacement Therapy (HRT) within the previous 6 months
* Subject has signs of acute or severe illness (i.e. unintentional weight loss, night sweats etc.)
* Subject has a known allergy or sensitivity to the investigational products or any ingredients of the investigational products
* Subject heavily consumes alcohol containing products defined as greater than (>) 3 drinks for men or 2 drinks for women (1 drink is 11 grams of alcohol or equivalence of 12 oz beer, 5 oz wine, or 1.5 oz distilled spirits) of alcoholic beverages per day
* Subject has donated more than 300 mL of blood during the last three months prior to screening
* Participating in another clinical trial
* Women who are premenopausal
* Subjects with active current psychiatric illness or condition which is likely to interfere with the subject's ability to understand the requirements of the biomedical research project
* Sunbed users will be excluded from the study.
* (Expected) increase in exposure to sunlight (e.g. a planned holiday of more than eight days, a beach holiday or a holiday outside Europe) in the study period of day 01 until day 28.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma 25(OH)D concentration at several visits | 6 months

SECONDARY OUTCOMES:
AUC(day1-day183) of 25(OH)D, 1,25(OH)2D, 24,25(OH)2D and vitamin D | 6 months
AUC(day1), Cmax(day1), Tmax(day1) and AUC(day182), Cmax(day182), Tmax(day182) of 25(OH)D, 1,25(OH)2D, 24,25(OH)2D and vitamin D | 6 months
Time point at which the plasma level of ≥75 nmol/L 25(OH)D is reached (t) | 6 months
Elimination rate and half-life of of 25(OH)D, 1,25(OH)2D, 24,25(OH)2D and vitamin D after cessation of supplementation | 6 months
Serum calcium and creatinine, albumin, PTH, urine calcium and creatinine and vital signs throughout the study, (Serious) Adverse event assessment and reporting | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hull, MSc, Principal Investigator — Leatherhead Food Research

REFERENCES:
- [Derived] Graeff-Armas LA, Bendik I, Kunz I, Schoop R, Hull S, Beck M. Supplemental 25-Hydroxycholecalciferol Is More Effective than Cholecalciferol in Raising Serum 25-Hydroxyvitamin D Concentrations in Older Adults. J Nutr. 2020 Jan 1;150(1):73-81. doi: 10.1093/jn/nxz209. PMID 31518424